CLINICAL TRIAL: NCT06848283
Title: Carotid Atherosclerosis Screening: Epidemiological Profile and Preventive Intervention
Brief Title: Randomized Controlled Trial on Carotid Atherosclerosis Screening in Asymptomatic Smokers and Hypertensive Adults: Prevalence and Impact on Cardiovascular Prevention
Acronym: CAROTID-CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CarotidAtheroScreening
Record Dates: First submitted 2025-02-12; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-12

CONDITIONS: Carotid Artery Atheroma; Cardiovascular Risk Stratification
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Ultrasonography, Carotid Arteries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Patients included in the intervention group will undergo a carotid ultrasonography (a non-invasive imaging exam) for the early detection of atherosclerotic plaques.
  Interventions: Diagnostic Test: Carotid ultrasonography
- Control Group (No Intervention): Control group (does not undergo carotid ultrasonography).

INTERVENTIONS:
Diagnostic Test: Carotid ultrasonography — All examinations will be performed by a technician specialized in neurosonology, using the same technical protocol. For this purpose, a portable ultrasound device with a linear probe (L3-9 MHz) will be used. A quick screening will be conducted to check for the presence of atherosclerosis.
  Arms: Intervention group

SUMMARY:
Title of the study: Carotid Atherosclerosis Screening: Epidemiological Profile and Preventive Intervention.

Objective: The main objective of this study is to characterize and identify the prevalence of carotid atherosclerosis in adults who are still asymptomatic for vascular disease and to evaluate the impact of detecting carotid atherosclerosis on preventive strategies. The study covers a population of approximately 4,780 patients.

Estimated Duration of the Project: The estimated duration of the project is 36 months, starting in February 2025, with the possibility of an extension if necessary.

Entities that approved the study: This study has been reviewed and approved by the Executive Director and President of the Clinical and Health Council of ACeS Grande Porto III - Maia/Valongo, as well as the Health Ethics Committee of the Northern Regional Health Administration (ARS Norte). The Addendum has also been approved by the Ethics Committee of the São João Local Health Unit (ULS São João).

Explanation of the Study:

This study will take place at ULS São João, including the São João University Hospital Center and the Primary Care Grouping (ACeS) Grande Porto III - Maia/Valongo.

The study includes two groups. Patients in the intervention group will undergo a neck ultrasound (a non-invasive imaging exam) for the early detection of atherosclerotic plaques. Demographic data (sex, age, educational level, employment status), vascular risk factors (smoking, alcohol consumption, blood pressure, and lipid profile), and anthropometric data (waist circumference and BMI) will be documented and analyzed by the research team. Medication, previous treatments, and other preventive initiatives will also be recorded. Glycemic and lipid profiles of participants will be collected.

Based on the results, the individual cardiovascular risk will be calculated using the SCORE2 global cardiovascular risk assessment chart from the European Society of Cardiology, both before and after incorporating ultrasound findings. Subsequently, personalized recommendations for preventive and therapeutic strategies will be developed for each patient and shared with family physicians.

To identify potential vascular risk biomarkers, venous blood samples will be collected in the intervention group. Patients identified with high-risk atherosclerotic plaques will be referred for further evaluation at the Neurology/Cerebrovascular Disease outpatient clinic of the São João University Hospital Center, ULS São João.

Patients in the other group (control group) will follow the same protocol, except for the neck ultrasound. To identify potential vascular risk biomarkers, venous blood collection will be performed in the intervention group during the carotid ultrasound (Doppler ultrasound). Both groups will be reassessed at a later stage. If a participant meets the exclusion criteria for the study, this will be duly explained to them.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥40 years and <70 years, hypertensive and smokers
* Registered in ACeS Maia/Valongo
* Willing to participate in the study

Exclusion Criteria:

* Inability to provide consent.
* Patients with a previous stroke, symptomatic coronary artery disease, or symptomatic peripheral artery disease will be excluded.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4780 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
To characterize and identify the prevalence of carotid atherosclerosis | From the beginning of the study until 2 years, with possible reassessments at intervals up to a maximum of 10 years.
  The main objective of this study is to characterize and identify the prevalence of carotid atherosclerosis in adults, smokers, and hypertensive individuals who are still asymptomatic for arterial vascular disease, and to evaluate the impact of having carotid atherosclerosis on preventive strategies.

SECONDARY OUTCOMES:
Describe the prevalence by severity of carotid atherosclerosis and relate it to vascular risk factors | From the beginning of the study until the reassessment after one year, with possible reassessments at intervals up to a maximum of 10 years.
  To describe the prevalence by severity of carotid atherosclerosis and relate it to sex, age, other known vascular risk factors (smoking, hypertension, diabetes, dyslipidemia, physical inactivity, alcohol consumption, overweight/obesity), and serum biomarkers; assess the potential protective effect of previous preventive treatments.
To evaluate the impact of carotid ultrasonography on cardiovascular risk | From the beginning of the study until the reassessment after one year, with possible reassessments at intervals up to a maximum of 10 years.
  To evaluate the impact of carotid ultrasonography on cardiovascular risk calculation and, consequently, on risk-adjusted preventive measures.
To assess the impact of carotid ultrasonography screening and the subsequent modifications in preventive measures on vascular events and mortality. | From the beginning of the study until the reassessment after one year, with possible reassessments at intervals up to a maximum of 10 years.
  The effects of preventive measures on the occurrence of vascular events (such as stroke and myocardial infarction), morbidity, and mortality rates will be reassessed one year after the initial evaluation.